CLINICAL TRIAL: NCT02076217
Title: Rates of Contraceptive Failure When Unprotected Intercourse Has Occurred 6-14 Days Prior to Contraceptive Initiation
Brief Title: Quick Start of Highly Effective Contraception
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Turok, MD, University of Utah
Other Study IDs: 67314
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: IUD; Contraceptive Implant; Contraception; Birth Control; Emergency Contraception
Keywords: Highly Effective Contraception; Emergency Contraception; Birth Control; LARC (Long Acting Reversible Contraception); HERC (Highly Effective Contraception)
MeSH Terms: interventions — Medroxyprogesterone Acetate; DEPO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (1):
- unprotected intercourse 6-14 days prior to contraception: Women who initiate highly effective reversible contraception within 6-14 days of unprotected intercourse.
  Interventions: Drug: Copper T-380 IUD; Drug: LNG IUD; Device: Contraceptive implant Nexplanon; Drug: Depo-Provera

INTERVENTIONS:
Drug: Copper T-380 IUD
  Other Names: Paragard IUD
Drug: LNG IUD
  Other Names: Mirena IUD, Skyla IUD
Device: Contraceptive implant Nexplanon
  Other Names: Etonorgestrel contraceptive implant, Implanon, Nexplanon
Drug: Depo-Provera
  Other Names: Depo, Intramuscular medroxyprogesterone acetate

SUMMARY:
This project will quantify rates of contraceptive failure when unprotected intercourse occurs 6-14 days prior to initiation of highly effective reversible contraceptives (such as IUD's and Implants).

DETAILED DESCRIPTION:
Women seeking emergency contraception (EC) frequently report multiple recent episodes of unprotected sex. Although high sensitivity urine pregnancy tests effectively rule-out pregnancy resulting from sex that occurred more than 14 days ago, clinicians are frequently concerned that pregnancy may result from unprotected sex that occurred <14 days prior to IUD placement. Placement of a copper IUD within 5 days of unprotected sex is a highly effective form of EC. Among 52 Chinese women who reported unprotected intercourse 5-7 days prior to copper IUD insertion, no pregnancies occurred. However, the effectiveness of the copper IUD when unprotected sex occurs 7-14 days prior to IUD placement is unknown. Intrauterine pregnancies rarely occur with a copper IUD in place. As some clinicians are concerned about injuring a pregnancy that occurs with an IUD in place, women who have had unprotected sex 7-14 days prior to requesting IUD placement are typically told they must use another, less effective, contraceptive for 2+ weeks and then return to obtain an IUD. To remove this barrier to emergency placement of a copper IUD, we propose to study rates of pregnancy when a copper IUD is placed "any time a urine pregnancy test is negative." We believe that simplifying guidance regarding the recommended timing of copper IUD placement has the potential to significantly increase the number of women offered "same-day" IUD service.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 15 and 45 years who request injectable, subdermal, or intrauterine contraception, 6-14 days after having unprotected intercourse.

Exclusion Criteria:

* History of tubal ligation or hysterectomy.
* Positive urine pregnancy test

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women presenting to IRB approved clinics requesting highly effective contraception (an IUD, Nexplanon®, or Depo-Provera) .
Sampling Method: Non-Probability Sample
Enrollment: 1030 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rates in the first month of contraceptive use | 4 weeks from contraception initiation
  This study is designed to provide clinicians and their patients with information regarding rates of contraceptive failure (i.e. undesired pregnancy) when contraception is initiated or placed for a woman who has a negative pregnancy test, but reports having had unprotected intercourse 6-14 days prior to requesting contraception.

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, Principal Investigator — University of Utah
Locations (1):
- Planned Parenthood Association of Utah, West Valley City, Utah, United States

REFERENCES:
- [Background] Sadler LS, Chen JY, Daley AM, Leventhal JM, Reynolds H. Reproductive care and rates of pregnancy in teenagers with negative pregnancy test results. J Adolesc Health. 2006 Mar;38(3):222-9. doi: 10.1016/j.jadohealth.2004.10.007. PMID 16488819
- [Background] Schwarz EB, Kavanaugh M, Douglas E, Dubowitz T, Creinin MD. Interest in intrauterine contraception among seekers of emergency contraception and pregnancy testing. Obstet Gynecol. 2009 Apr;113(4):833-839. doi: 10.1097/AOG.0b013e31819c856c. PMID 19305327
- [Background] Westhoff C, Kerns J, Morroni C, Cushman LF, Tiezzi L, Murphy PA. Quick start: novel oral contraceptive initiation method. Contraception. 2002 Sep;66(3):141-5. doi: 10.1016/s0010-7824(02)00351-7. PMID 12384200
- [Derived] Boraas CM, Sanders JN, Schwarz EB, Thompson I, Turok DK. Risk of Pregnancy With Levonorgestrel-Releasing Intrauterine System Placement 6-14 Days After Unprotected Sexual Intercourse. Obstet Gynecol. 2021 Apr 1;137(4):623-625. doi: 10.1097/AOG.0000000000004118. PMID 33706343